CLINICAL TRIAL: NCT00371332
Title: Effect of Adjunctive Treatment With Arestin on the Subgingival Microflora in Patients With Moderate to Advanced Periodontitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: OraPharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OPI-145'
Record Dates: First submitted 2006-09-01; First posted 2006-09-04 (Estimated); Last update posted 2006-09-25 (Estimated); Status verified 2006-09

CONDITIONS: Periodontitis
Keywords: chronic periodontitis, mouth; Moderate to advanced chronic periodontitis
MeSH Terms: conditions — Periodontitis; Chronic Periodontitis

INTERVENTIONS:
Drug: Minocycline HCL Microspheres

SUMMARY:
The purpose of this study is to measure the antimicrobial effects of Arestin in subjects with moderate to advanced periodontal disease

ELIGIBILITY:
Inclusion Criteria:

* Generalized moderate to advanced chronic periodontitis, five sites with probing depths of >5 mm in 5 non-adjacent interproximal spaces, excluding the distal of terminal teeth, at least 16 teeth excluding 3rd molars and implants

Exclusion Criteria:

* Allergy to tetracycline
* Subjects with aggressive periodontitis
* Acute necrotizing ulcerative gingivitis, or gross decay
* Systemic conditions which could influence the course of periodontal disease (i.e, diabetes, autoimmune disease, etc)
* Individuals requiring prophylactic antibiotics
* Any periodontal therapy within the previous 3 months (excluding maintenance therapy)
* Systemic or local antibiotic therapy within three months

Ages: 30 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 128
Dates: Start 2004-01

PRIMARY OUTCOMES:
The change in the mean sum of primary pathogens (P. gingivalis, To forsythensis, and T. denticola) from baseline to 30 days.

SECONDARY OUTCOMES:
Changes in the numbers of each of the primary pathogens, changes in pocket depth, attachment level, and proportion of sites bleeding on probing

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Los Angeles, California
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Buffalo, New York
  - Memphis, Tennessee

REFERENCES:
- See also: Effect of Adjunctive Treatment with Arestin on the Subgingival Microflora in Patients with Moderate to Advanced Periodontitis — http://download.veritasmedicine.com/PDF/OPI-145_CSR.pdf